CLINICAL TRIAL: NCT02716974
Title: A Phase II Study of Definitive Therapy for Newly Diagnosed Men With Oligometastatic Prostate Cancer
Brief Title: A Study of Definitive Therapy to Treat Prostate Cancer
Acronym: oligo-mets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1618; IRB00070003 (Other: JHM IRB)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
Keywords: Lupron; Bicalutamide; Docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; bicalutamide; Docetaxel; Prostatectomy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemohormonal and definitive therapy (Experimental): (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of neoadjuvant androgen deprivation (Leuprolide Acetate) and up to 6 cycles of chemotherapy (Docetaxel), (2nd) definitive local tumor control with prostatectomy +/- adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. The men will receive a total of 1 year of androgen deprivation. Androgen blockade (Bicalutamide) will be the same throughout the course of treatment.
  Interventions: Drug: Leuprolide Acetate; Drug: Bicalutamide; Drug: Docetaxel; Procedure: Prostatectomy; Radiation: Radiation

INTERVENTIONS:
Drug: Leuprolide Acetate — 22.5mg by intramuscular (IM) injection every 3 months
  Other Names: Lupron Deport
Drug: Bicalutamide — bicalutamide (Casodex) 50mg by mouth daily
  Other Names: Casodex
Drug: Docetaxel — Docetaxel (taxotere) 75 mg/m2 IV will be given on day 1 every 3 weeks, up to 6 cycles.
  Other Names: Texotere
Procedure: Prostatectomy — Removal of the entire prostate gland, plus some surrounding tissue.
  Other Names: Radical prostatectomy
Radiation: Radiation — 5 high dose radiation treatments to the metastatic (tumor has spread to other parts of the body) sites.

SUMMARY:
To assess the safety of treating men with oligometastatic prostate cancer with the following therapy: (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of neoadjuvant androgen deprivation and up to 6 cycles of chemotherapy, (2nd) definitive local tumor control with prostatectomy +/- adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. The men will receive a total of 1 year of androgen deprivation. Androgen blockade will be the same throughout the course of treatment.

DETAILED DESCRIPTION:
Neoadjuvant treatment (month 1 through ~6): All patients will be treated with up to 6 months of androgen deprivation, plus up to 6 cycles of docetaxel chemotherapy. Following docetaxel therapy, patients with a prostate-specific antigen response of at least a 50% decrease from baseline, will proceed to maximum consolidative therapy.

Surgery and Radiation (month 7 though ~11): After completion of neoadjuvant therapy, the men will be treated with definitive local therapy with radical prostatectomy (RP) +/- adjuvant radiation therapy (RT). After definitive local therapy, patients will be treated with consolidative stereotactic body radiation therapy (SBRT) to the metastatic sites.

Follow up: Patients will continue on androgen deprivation for a total of 1 year. They will be followed clinically and monitored with serum testosterone and prostate-specific antigen until 2-years after completion of ADT (Androgen deprivation therapy) treatment. Androgen blockade will be the same throughout the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Age ≥ 18 years
* Eastern cooperative group (ECOG) performance status ≤2
* Documented histologically confirmed adenocarcinoma of the prostate
* Willing to undergo the following therapy: (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of neoadjuvant androgen deprivation and up to 6 cycles of chemotherapy, (2nd) definitive local tumor control with prostatectomy +/- adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. Additionally, must be willing to be treated with a full year of androgen deprivation.
* Oligometastatic prostate cancer: Stage T1-4, N0-1 and/or M1a-b (up to 5 metastatic lesions- including bone lesions and non-regional lymph nodes seen on bone scan, contrast enhanced CT scan, or positron emission tomography scan)
* Able to swallow the study drugs whole as tablets

Exclusion Criteria:

* Prior local therapy to treat prostate cancer (e.g. radical prostatectomy, radiation therapy, brachytherapy)
* Prior therapy to a metastatic site.
* Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

  1. Hormonal therapy (e.g. leuprolide, goserelin, triptorelin, degarelix)
  2. Cytochrome (CYP) -17 inhibitors (e.g. ketoconazole)
  3. Antiandrogens (e.g. bicalutamide, nilutamide)
  4. Second generation antiandrogens (e.g. enzalutamide, abiraterone)
  5. Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  6. Chemotherapy (e.g. docetaxel, cabazitaxel) *Note: may be enrolled if hormone therapy was recently initiated (<90 days duration). In the event that hormone therapy was initiated prior to study enrollment, the clock for 1 year of androgen deprivation would begin at the time of therapy initiation, rather than at study enrollment.
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
* Abnormal bone marrow function [absolute neutrophil count (ANC)<1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL]
* Abnormal liver function (bilirubin >upper limit of normal; aspartate aminotransferase , alanine aminotransferase > 2.5 x upper limit of normal)
* Creatinine clearance of ≥ 30 mL/min. Creatinine clearance should be calculated suing the Cockcroft-Gault formula.
* Active cardiac disease defined as active angina, symptomatic congestive heart failure, or myocardial infarction within previous six months.
* Prior history of malignancy in the past 3 years with the exception of basal cell and squamous cell carcinoma of the skin. Other malignancies that are considered to have a low potential to progress may be enrolled at discretion of PI.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pienta, MD, Principal Investigator — SKCCC at Johns Hopkins University
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemohormonal and Definitive Therapy
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemohormonal and Definitive Therapy
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 59.8 [55.1 to 69.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed by 2-year PSA Progression-free Survival Rate
Description: To evaluate efficacy of multimodality therapy in men, defined as the 2 year PSA progression-free (PSA<0.2 ng/ml) survival among men who have non-castrate testosterone levels 2 years after enrollment. Number of participants (who have non-castrate testosterone levels 2 years after enrollment) with PSA progression-free survival.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemohormonal and Definitive Therapy
Number analyzed (Participants) | 26
Participants | 17

2. Secondary Outcome: Safety of the Multimodality Therapy as Assessed by Number of Participants With Neutropenia and Surgical or Radiation Toxicities
Description: To assess the safety and therapeutic benefit of multimodality therapy in men presenting with newly diagnosed oligometastatic prostate cancer (<5 sites of metastases). Safety is defined as the incidence of Grades 3 and 4 neutropenia and surgical- or radiation-induced toxicities.
  Neutropenia is a lower than normal number of neutrophils (a type of white blood cell) in the blood. Although dependent on the specific laboratory, the normal number is of neutrophils is generally about 1500-7800 cells/microliter. Grade 3 and 4 neutropenia refer to neutrophil levels <1,000-500 and <500, respectively. The average risk of docetaxel-induced Grade 3 and 4 neutropenia is about 35%. During the course of the study, if we had seen evidence that the risk of Grade 3 and 4 neutropenia was >50%, the study would have been stopped.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Chemohormonal and Definitive Therapy
Number analyzed (Participants) | 26
Participants | 26

3. Secondary Outcome: Time to Prostate-specific Antigen Recurrence
Description: To investigate the time from an undetectable prostate-specific antigen (≤0.2 ng/mL) until the prostate-specific antigen is >0.2 over two time-points.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemohormonal and Definitive Therapy
Number analyzed (Participants) | 26
Months | 31 [25.2 to 32.3]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Chemohormonal and Definitive Therapy
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemohormonal and Definitive Therapy (N=26)
back pain (Injury, poisoning and procedural complications) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
partial bowel obstruction (Gastrointestinal disorders) | 1 (1)
neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemohormonal and Definitive Therapy (N=26)
edema (General disorders) | 5 (6)
alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 2 (2)
urinary incontinence (Renal and urinary disorders) | 3 (4)
bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 2 (2)
nerve pain (Nervous system disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 15 (15)
hot flashes (Vascular disorders) | 11 (11)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
headache (Nervous system disorders) | 2 (2)
muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 2 (2)
dysgeusia (Nervous system disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 4 (5)
neuropathy (Nervous system disorders) | 6 (7)
anemia (Blood and lymphatic system disorders) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
white blood cell decreased (Blood and lymphatic system disorders) | 3 (4)
blurred vision (Eye disorders) | 1 (1)
insomnia (Psychiatric disorders) | 3 (3)
alkaline phosphatase increased (Investigations) | 1 (1)
xerostomia (Gastrointestinal disorders) | 2 (3)
pruritus (Infections and infestations) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
weight gain (Investigations) | 1 (1)
hypertension (Vascular disorders) | 1 (3)
bilirubin increased (Hepatobiliary disorders) | 1 (1)
(Serum Glutamic-Oxaloacetic Transaminase)SGOT increased (Investigations) | 1 (2)
(Serum Glutamic-Pyruvic Transaminase) SGPT increased (Investigations) | 1 (1)
infusion reaction (General disorders) | 1 (2)
floater eyes (Eye disorders) | 1 (1)
decreased libido (Psychiatric disorders) | 1 (1)
neutrophil count decreased (Blood and lymphatic system disorders) | 1 (2)
lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
stress incontinence (Psychiatric disorders) | 2 (2)
intermittent dizziness (Nervous system disorders) | 1 (1)
metallic taste (Nervous system disorders) | 1 (1)
flushed face (Skin and subcutaneous tissue disorders) | 1 (1)
right arm rash (Skin and subcutaneous tissue disorders) | 1 (1)
(GERD)gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02716974/Prot_SAP_000.pdf